CLINICAL TRIAL: NCT05412368
Title: Enhancing CAMHS Referrals: EnCAMHS
Brief Title: Enhancing Referrals to Child and Adolescent Mental Health Services: EnCAMHS
Acronym: EnCAMHS
Status: Completed | Type: Observational
Sponsor: Greater Manchester Mental Health NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other); Manchester University NHS Foundation Trust (Other Government); Pennine Care NHS Foundation Trust (Other Government); Northumberland, Tyne and Wear NHS Foundation Trust (Other); MQ Mental Health (Unknown); Anna Freud National Centre for Children and Families (Other); McPin Foundation (Other); 42nd Street (Unknown)
Responsible Party: Principal Investigator, Kathryn Abel, Professor Kathryn Abel, Greater Manchester Mental Health NHS Foundation Trust
Other Study IDs: NIHR131379
Record Dates: First submitted 2022-04-28; First posted 2022-06-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Mental Health Issue
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children and young people (CYP): Children and young people who have been referred to CAMHS
  Interventions: Other: Focus Groups
- Parents/carers: Parents/carers of CYP who have been referred to CAMHS
  Interventions: Other: Focus Groups
- Key referrers: Key referrers (e.g. Teachers, GPs, SENCOs, Social Workers) who have referred CYP to CAMHS
  Interventions: Other: Focus Groups
- CAMHS Professionals: CAMHS Professionals who have received referrals to CAMHS
  Interventions: Other: Focus Groups

INTERVENTIONS:
Other: Focus Groups — Focus Groups

SUMMARY:
Our aim is to find low-cost and widely reusable mechanisms to reduce inappropriate referrals. Our key objectives are:

Engage with key stakeholders to identify problems with making appropriate referrals Analyse CAMHS referral data to understand and identify problems (quantitatively) Identify requirements for sustainable solutions Explore with key stakeholders how we can improve the referral process Identify how the best proposed solutions could be embedded within routine CAMHS referral pathways

DETAILED DESCRIPTION:
The Investigators shall conduct a series of focus groups with key stakeholders involved in the referral to CAMHS process; children and young people (CYP), parents/carers, key referrers, CAMHS professionals in order to better understand the challenges that exist with the current referral process. Following this, the Investigators will conduct further focus groups with the key stakeholders above, in which they will suggest sustainable solutions to the problems that have been identified.

The Investigators shall then identify how the propose solutions can be embedded into routine CAMHS referral pathways.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years and above
* have experience of CAMHS referral pathway

Exclusion Criteria:

* younger than 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anyone aged 16 and above who has been involved in the CAMHS referral pathway
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Solutions to enhance the referral process for CAMHS | By end of study - within 1 year
  Solutions to help improve the referrals into CAMHS, using data collected during focus groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We will not be sharing IPD

REFERENCES:
- [Derived] Abel KM, Whelan P, Carter LA, Tranter H, Stockton-Powdrell C, Gutridge K, Hassan L, Elvins R, Edbrooke-Childs J. Enhancing referrals to Child and Adolescent Mental Health Services: the EN-CAMHS mixed-methods study. Health Soc Care Deliv Res. 2025 Jun;13(21):1-59. doi: 10.3310/GYDW4507. PMID 40521776